CLINICAL TRIAL: NCT05125601
Title: Hearing Quality of Life of Children With Hearing Aids: Study Based on the PEACH Questionnaire
Brief Title: PEACH Questionnaire Study
Acronym: QaPEACH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211111; 2021-A01468-33 (Other: ID RCB number)
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Deafness
Keywords: Deafness in children; The Parents' Evaluation of Aural/Oral Performance of Children (PEACH) in french
MeSH Terms: conditions — Deafness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with bilateral deafness: Patients aged 2 to 10 years with bilateral deafness, wearing an amplifier device and / or a cochlear implant.
  Interventions: Other: The Parents' Evaluation of Aural/Oral Performance of Children (PEACH)

INTERVENTIONS:
Other: The Parents' Evaluation of Aural/Oral Performance of Children (PEACH) — The Parents' Evaluation of Aural/Oral Performance of Children (PEACH) will be completed once.
  Other Names: Questionnaire

SUMMARY:
There are few or no questionnaires in French on the hearing quality of life of children with hearing aids.

The objectives of the study are to measure the hearing quality of life of children with hearing aid and / or cochlear implants and to compare the hearing quality of life according to the type of hearing aid (hearing aid and / or cochlear implant).

DETAILED DESCRIPTION:
There are few or no questionnaires in French on the hearing quality of life of children with hearing aids.

The study will allow an evaluation of the quality of life benefit of hearing rehabilitation at different ages and with varying levels of deafness.

The translated questionnaire for the study will be given to the parents of the child after a sure diagnosis of the child's degree of deafness and at least 1 month of hearing aids. The translated is proposed by Necker Hospital Pediatric ENT department.

The objectives of the study are to measure the hearing quality of life of children with hearing aid and / or cochlear implants and to compare the hearing quality of life according to the type of hearing aid (hearing aid and / or cochlear implant).

ELIGIBILITY:
Inclusion Criteria:

* Minors aged 2 to 10 years (inclusive)
* Patients followed in consultation at Necker Hospital in the Pediatric ENT department
* With a slight to deep bilateral deafness
* Auditory experience with hearing aid and / or cochlear implant bilateral for more than 1 month
* holders of parental authority not opposed to participation in the study

Exclusion Criteria:

* Non-wearing of hearing aid and / or implant over the last month
* malfunction of hearing aids and / or implant
* Non-understanding of the French language by parents

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients followed by the Pediatric ENT department of Necker-Enfants Malades hospital.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Hearing quality of life | Day 0
  Score at the Peach questionnaire: qualitative assessment of the perception with the equipment in various modalities of everyday life.
  The Peach questionnaire is composed of 13 questions with the possibility of setting a score between 0 (never) and 4 (always). Each questionnaire gives an average of the embarrassment of the children in the silence and in the noise. The results will give the opportunity to change the settings, evaluate the quality of the hearing aid and the change them if it is necessary.

SECONDARY OUTCOMES:
Difference of score to the Peach questionnaire according to the type of hearing aids | Day 0
  Difference of scores according to the hearing aid:
  * Bilateral hearing aid,
  * Bilateral cochlear implant,
  * A cochlear implant on one side and an auditory device on the other. The Peach questionnaire is composed of 13 questions with the possibility of setting a score between 0 (never) and 4 (always). Each questionnaire gives an average of the embarrassment of the children in the silence and in the noise. The results will give the opportunity to change the settings, evaluate the quality of the hearing aid and the change them if it is necessary.
Difference of score to the Peach questionnaire according to the type of deafness | Day 0
  Difference of scores according to the degree of deafness as well as the origin of deafness: congenital non-evolutive, evolutive.
  The Peach questionnaire is composed of 13 questions with the possibility of setting a score between 0 (never) and 4 (always). Each questionnaire gives an average of the embarrassment of the children in the silence and in the noise. The results will give the opportunity to change the settings, evaluate the quality of the hearing aid and the change them if it is necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie LOUNDON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Tabatha DERAY, Hearing Care Professional, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No